CLINICAL TRIAL: NCT02904681
Title: Multicenter Retrospective Evaluation of the Surgical Management of Spinal Growth Dystrophy
Acronym: DRC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DRC
Record Dates: First submitted 2016-08-31; First posted 2016-09-19 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Acetabular Fractures; Hip Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention. Observational and descriptive study

SUMMARY:
Spinal growth dystrophy (CRD), also called Scheuermann's disease, corresponding to impaired vertebral structure occurring in children and adolescents with involvement of the growth cartilage causing impaired growth and kyphosis.

There are forms thoracolumbar and thoracic conventional forms of DRC with variable clinical expressions; the most important being kyphosis with spinal stiffness associated with painful elements.

The radiographic definition according Sorenson is uniformisation 5 ° affecting at least three adjacent vertebrae.

Scheuermann's disease and three problems. First, the thoracic kyphosis generates back pain which may be thoracic or lumbar indirectly attributed to compensatory lordosis. Moreover disruption sagittal balance frequently causes a significant aesthetic discomfort. Finally, scalability because the curvature may increase the likelihood of degenerative lesions disc degeneration or lumbar spinal stenosis for example.

When the disease is diagnosed early, treatment is most often associated with orthopedic physiotherapy. However, for patients with active deformation, despite an orthopedic brace treatment with chronic pain, neurological deficit or for aesthetic reasons, surgical decision can be taken.

The goal of surgical treatment of DRC is a correction of the thoracic kyphosis. It goes through a spinal fusion must be released from his column stiffness in a bad position, changing the equilibrium profile and ensure that it remains in a good position.

This surgery usually requires a prior operative time (thoracic surgery to remove the intervertebral discs) and a posterior surgical time (blockage of the vertebrae together with a bone graft and osteosynthesis). Currently different surgical strategies are practiced there is no real consensus between the teams.

DETAILED DESCRIPTION:
objectives:

1. Evaluation of the rate and type of complications in different age categories and surgical strategies.
2. Evaluation of clinical results based on surgical strategies.
3. Evaluation of sagittal balance and correction obtained based surgical strategies

Methodology and duration of the research

This is a multicenter retrospective cohort on the assessment of surgical practices cited objectives. Also, this research is in Chapter X of the Data Protection Act and allows the collection of personal data for the purpose of evaluation of care and prevention practices with authorization request to the CNIL; the opinion of CCTIRS therefore not required in this case.

This study concerns the data of patients operated with the techniques mentioned in addition with a decline of more than 20 years.

Patients are aware of the potential use of their data in their files for medical research through oral information provided by the doctor at the signing by the patient's consent related to the surgery and most recently contained in the Home booklet setting for patients.

Nature of the data collected

The data is anonymous and not identifiable (for each subject a number of inclusion is given). The name of the surgeon is also anonymized.

The data collected concern the characteristics of the patient, as well as its history, the operating data including technical, suites and possible post-operative complications and patient monitoring.

Data collection will be done on the basis KEOPS https://www.keops-spine.fr

ELIGIBILITY:
Inclusion Criteria:

* patients operated on for an arthrodesis Dystrophy Spinal Growth (DRC)
* Age> 10 years
* monitoring of minimum one year

Exclusion Criteria:

* deformation in the frontal plane
* kyphosis malformation
* osteoporotic or degenerative kyphosis
* post laminectomy kyphosis
* constitutional bone disease
* connective Tissue Disease
* myopathy

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated on for an arthrodesis Dystrophy Spinal Growth (DRC)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
Surgery complication type | Day 30
  Statement from the database keops

SECONDARY OUTCOMES:
Assessment od the clinical results based on surgical strategies | Day 30
  Evaluation of clinical results based on surgical strategies. Statement from the database keops :
  * Worse,
  * Acceptable,
  * Good
Assessment of sagittal balance and correction Score obtained | Day 30
  Evaluation of sagittal balance score obtained based surgical strategies. Statement from the database keops:
  * Worse,
  * Acceptable,
  * Good
Assessment of correction Score obtained | Day 30
  Evaluation of sagittal correction score obtained based surgical strategies. Statement from the database keops:
  * Worse,
  * Acceptable,
  * Good

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided